CLINICAL TRIAL: NCT07250256
Title: Radiographic and Histomorphometric Evaluation of Xenograft as a Socket Preservation Material in Maxillary Posterior Teeth: A Randomized-Controlled Clinical Study
Brief Title: Radiographic and Histomorphometric Evaluation of Xenograft as a Socket Preservation Material in Maxillary Posterior Teeth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 547-2022
Record Dates: First submitted 2025-08-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Socket Preservation
Keywords: Socket; Healing; bone formation; histomorphometery

STUDY DESIGN:
Intervention Model Description: This is an In-Vivo comparative randomized controlled study that will be conducted on patients of the outpatient clinic of Oral and Maxillofacial department Suez Canal University to evaluate the difference between using S1-XB bone graft as a socket preservation material and normal socket healing without adding any socket preservation materials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): (8 cases): was treated by immediate socket preservation with S1-XB xenograft augmentation after extraction.
  Interventions: Device: S1-XB
- Control group (Placebo Comparator): (8 cases): was not exposed to any type of socket preservation after the extraction procedure.
  Interventions: Procedure: Control (Standard treatment)

INTERVENTIONS:
Device: S1-XB — Socket grafted with xenograft containing alginate hydrogel material
  Arms: Study group
Procedure: Control (Standard treatment) — Atraumatic extraction and sockets were allowed to undergo normal healing without any graft materials
  Arms: Control group

SUMMARY:
Radiographic and Histomorphometric Evaluation of Xenograft as a Socket Preservation Material in Maxillary Posterior Teeth: A Randomized-Controlled Clinical Study

DETAILED DESCRIPTION:
The process of natural healing starts with new bone formation taking place from initial islands of bone within the connective tissue occurring after a 4 to 8 weeks interval from extraction date. This is followed by the manifestation of a mature trabecular structure that can be noticed at 10 to 20 weeks after extraction accompanied with a reduction in osteoblast count. As a result of the extensive bone resorption post extraction, the prosthetically driven implant placement is compromised and in need of some ridge preservation techniques that have been widely studied to try and ensure less alveolar bone loss. The aim of this research is to study the S1-XB Xenograft containing hydrogel and to evaluate its effects on extraction socket healing in comparison to natural socket healing. This is an In-Vivo comparative randomized controlled study that will be conducted on patients of the outpatient clinic of Oral and Maxillofacial department Suez Canal University to evaluate the difference between using S1-XB bone graft as a socket preservation material and normal socket healing without adding any socket preservation materials.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged between 21 and 40 years.
* General good health.
* Absence of any relevant systemic disease.
* Presence of a hopeless maxillary posterior tooth that requires extraction.
* Extraction site suitable for replacement by a dental implant.
* Cases have adequate bone width and length.
* Volunteer subjects must sign an informed consent.

Exclusion Criteria:

* Poor oral hygiene with no possibility of improvement.
* Smokers (more than 10 cigarettes per day).
* Chronic treatment with any medication known to affect oral status and bone turnover.
* Drug or alcohol abuse.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — males with general good health. Non smokers
Enrollment: 16 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Histomorphometric analysis | 16 weeks
  Samples were first stained with hematoxylin and eosin (H&E) to demonstrate the general tissue architecture, cellular distribution, and overall structural organization. Subsequently, sections were stained with Masson's Trichrome (MTC) to allow both qualitative and quantitative assessment of bone trabeculae and osteoid tissue. Osteopontin (OPN) immunohistochemistry was used to assess the percentage of OPN expression area within the surrounding connective tissue. The OPN poly-colonal antibody was purchased from Thermo Fisher Scientific, Catalog # PA1-72061. Images were captured at ×400 magnification using a SOPTOP EX20 microscope with HD camera. ImageJ software was used to quantify area% from five standardized fields per section at oral pathology laboratory, Faculty of Dentistry, Suez Canal University.
Radiographic evaluation | 16 weeks
  Cone-beam computed tomography (CBCT) scans (Scanora 3D) were obtained immediately after extraction at baseline and postponed at 4 months postoperatively to evaluate the following parameters: bone density that was measured in Hounsfield units (HU) at the center of the socket, ridge height that was determined by vertical distance from the crestal bone to a fixed reference point and ridge width that was measured at 3 mm apical to the crest.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal university, Ismailia, Egypt